CLINICAL TRIAL: NCT03086434
Title: Intertribal Talking Circle for the Prevention of Substance Abuse in Native Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Northern Arizona University (Other); Choctaw Nation of Oklahoma (Unknown); University of North Carolina (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017.19687
Record Dates: First submitted 2017-03-02; First posted 2017-03-22 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2018-08

CONDITIONS: Substance Use
Keywords: Culturally tailored intervention; American Indian early adolescents; Prevention of substance use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally tailored intervention (Experimental): The participants of the experimental condition will receive the intervention in a talking circle format. They will meet for 10 weekly 50 minute sessions.
  Interventions: Other: Culturally Tailored Intervention
- Standard Substance Abuse Education (Active Comparator): The control condition participants are assigned to the standard substance abuse education program which is delivered in a classroom format format. They will meet for 10 weekly 50 minute classroom sessions.
  Interventions: Other: Standard Substance Abuse Education

INTERVENTIONS:
Other: Culturally Tailored Intervention — School-based substance use prevention
  Arms: Culturally tailored intervention
Other: Standard Substance Abuse Education — Class room program
  Arms: Standard Substance Abuse Education

SUMMARY:
This project will evaluate an after-school substance abuse prevention intervention, compared to a standard substance abuse education program, targeting 6th grade AI youth in three AI communities: Ojibwe/Chippewa in Minnesota, Choctaw in Oklahoma, and Lumbee in North Carolina.

A community-based participatory research approach will be used to culturally and technologically adapt the intervention. A two-condition controlled study will evaluate the efficacy of the intervention to increase AI youth Native self-reliance while decreasing AI youth substance use involvement. An adult training program second level intervention study will also be implemented to train tribal personnel from the three regional tribes on how to implement the intervention as a tribal program beyond the study period.

Effectiveness will be determined by a small partial cross-over randomized trial comparing the intervention to a wait-list control condition. Process evaluations will focus on the future adoption and implementation of the intervention, and recommendations for sustainable adaptations.

DETAILED DESCRIPTION:
The proposed study will consist of a 5-year plan: Year 1 has been completed and consisted of strengthening and extending community partnerships in each community and collecting data that will inform the cultural adaptation and tailoring of the intervention; Years 2, 3, and 4 will entail implementation by using a two-condition controlled study in which the culturally competent intervention is compared to standard care; and Year 5 will consist of final data collection, analysis of results, dissemination of results to local communities, and finalization of a sustainability plan for each Tribe.

Participants in the proposed study will consist of 540 male and female American Indian 6th grade students who represent at least three different Tribes - Choctaw, Ojibwe/ Chippewa, and Lumbee, in three different regions of the U.S. Participants will also include 70 tribal personnel (adults 18 and over) who be trained to implement the intervention in Years 3 & 4 of the project. Finally, 15-20 stakeholders and community partnership members will be interviewed at various stages of this project.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for youth participants include:
* AIl students enrolled in the 6th grade at each of the 3 regions
* Active parental consent
* Student willingness to participate and signed assent. Inclusion criteria for adult participants include: adults over 18 years of age currently employed as personnel, educators, and counselors at tribal schools among the three regions.

Exclusion Criteria:

* Exclusion criteria include students who are not identified as American Indian, no active parental consent, and no signed assent.

Ages: 10 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 630 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
Substance Use | Change overtime at baseline, 6 months, 12 months
  Self-report to substance use

SECONDARY OUTCOMES:
Native Self-Reliance | Change overtime at baseline, 6 months, 12 months
  Cultural identity

CONTACTS AND LOCATIONS:
Overall Officials: John Lowe, PhD, Principal Investigator — Florida State University

IPD SHARING:
Plan to Share IPD: Yes
This study and project will be presented to the other researchers and at national conferences and submitted for publication after study completion.